#### MEDICAL RECORD

#### CONSENT TO PARTICIPATE IN A CLINICAL RESEARCH STUDY

Adult Patient or

• Parent, for Minor Patient

INSTITUTE: National Cancer Institute

STUDY NUMBER: 10-C-0011 PRINCIPAL INVESTIGATOR: Wyndham H. Wilson, M.D., Ph.D.

STUDY TITLE: Phase II Trial of Alemtuzumab (Campath) and Dose-Adjusted EPOCH-Rituximab (DA-

EPOCH-R) in Relapsed or Refractory Diffuse Large B-Cell and Hodgkin Lymphomas

Continuing Review Approved by the IRB on 09/24/18

Amendment Approved by the IRB on 09/04/18 (J)

Date posted to web: 10/06/18

Standard

#### INTRODUCTION

We invite you to take part in a research study at the National Institutes of Health (NIH).

First, we want you to know that:

Taking part in NIH research is entirely voluntary.

You may choose not to take part, or you may withdraw from the study at any time. In either case, you will not lose any benefits to which you are otherwise entitled. However, to receive care at the NIH, you must be taking part in a study or be under evaluation for study participation.

You may receive no benefit from taking part. The research may give us knowledge that may help people in the future.

Second, some people have personal, religious or ethical beliefs that may limit the kinds of medical or research treatments they would want to receive (such as blood transfusions). If you have such beliefs, please discuss them with your NIH doctors or research team before you agree to the study.

Now we will describe this research study. Before you decide to take part, please take as much time as you need to ask any questions and discuss this study with anyone at NIH, or with family, friends or your personal physician or other health professional.

# Why is this study being done?

The general purpose of this study is to develop treatments for lymphoma that are more effective than existing therapies. The experimental part of this treatment program is to test whether giving campath (alemtuzumab) in combination with continuous infusion EPOCH-rituximab chemotherapy will improve the outcome of therapy of your lymphoma. In this study five chemotherapy drugs are given together in an intensive combination called EPOCH. In addition, you will receive a drug called rituximab. EPOCH-R contains drugs which are standard for the treatment of lymphomas. Because higher doses of chemotherapy may increase the benefit, the doses of several drugs in EPOCH-R may be increased on each cycle if you tolerated them on the previous cycle.

PATIENT IDENTIFICATION

#### CONSENT TO PARTICIPATE IN A CLINICAL RESEARCH STUDY

• Adult Patient or Parent, for Minor Patient NIH-2514-1 (07-09)

P.A.: 09-25-0099

| Study | MEDICAL RECORD | CONTINUATION SHEET for either: NIH 2514-1, Consent to Participate in A Clinical Research Study NIH 2514-2, Minor Patient's Assent to Participate In A Clinical Research Study |
|---|---|---|
|---|---|---|

STUDY NUMBER: 10-C-0011 CONTINUATION:  pages

# Why are you being asked to take part in this study?

You have a disease called Diffuse Large B-cell lymphoma or Hodgkin lymphoma which your doctors think would be best treated with chemotherapy. This protocol is specifically for people with diffuse large B-cell or Hodgkin lymphomas, as we are trying to find better treatments for these types of lymphoma.

# How many people will take part in this study?

Approximately 52 subjects will participate in this study.

# **Description of Research Study**

Studies conducted at the National Cancer Institute suggest that certain chemotherapy drugs may be more effective if given by continuous infusion into the vein rather than by the standard method of rapid intravenous injection. One such combination, which we call EPOCH (each letter stands for one of the drugs used in the combination), seems to have a high degree of effectiveness in patients whose tumors have stopped responding to standard regimens. Recent evidence also indicates that the effects of chemotherapy may be improved by combination with monoclonal antibodies. Monoclonal antibodies are purified proteins that are specially made to attach to pieces of foreign substances (such as cancer cells) with the goal of inactivating them. A monoclonal antibody, called campath (Alemtuzumab), has been manufactured to attach to a protein called CD52 that may target your tumor cells or the surrounding inflammatory cells. Rituximab is another monoclonal antibody that you will receive which binds to a specific molecule (called CD20) present on most B-cells and is part of standard therapy. We performed a study using the combination of EPOCH and campath in other types of lymphomas. Based on this previous study, we have experience with this combination of drugs, especially with regards to its safety and the optimal doses of the drug used. Most patients experienced mild infusional reactions, manifesting as fever, chills and rash. Documented infections were common and the most common were viral infections. The most common virus detected was cytomegalovirus which generally did not produce symptoms and is detected only by a blood test. Other types of infections seen were bacterial and fungal infections but these occurred less frequently. Based on positive results we have had in the past treating lymphomas with EPOCH combined with rituximab or campath, we now plan to test this combination of EPOCH-RC in patients who have previously been treated with chemotherapy and have either relapsed or are refractory to the prior chemotherapy regimen. Up to 52 patients will be treated on this study. All of the drugs used in this protocol have been FDA approved.

# What will happen if you take part in this research study?

#### Before you begin the study

In order to determine if you are eligible for this study, several tests need to be done. This period of evaluation may take up to three weeks and may be done on an outpatient basis. Evaluation may include some or all of the following tests: standard blood tests, 24 hour collections of urine, tests of lung and heart function, computerized tomography (CT) scans, nuclear medicine scans of the body (called a PET scan), bone marrow biopsies and biopsies of suspected areas of tumor.

#### PATIENT IDENTIFICATION CONTINUATION SHEET for either:

NIH-2514-1 (07-09) NIH-2514-2 (10-84) P.A.: 09-25-0099

| MEDICAL RECORD | CONTINUATION SHEET for either: NIH 2514-1, Consent to Participate in A Clinical Research Study NIH 2514-2, Minor Patient's Assent to Participate In A Clinical Research Study |
|---|---|
|---|---|

STUDY NUMBER: 10-C-0011 CONTINUATION:  pages

#### **During the study**

EPOCH-R-Campath chemotherapy treatment: The chemotherapy regimen known as EPOCH-RC will be given by intravenous (IV) infusion through a "central line," an IV catheter (or tube) placed in a large vein in your arm or chest. You will be admitted to the hospital for the infusion of the monoclonal antibody therapy on this protocol but may receive the chemotherapy infusion as an outpatient. Patients will receive dose adjusted (DA) EPOCH-R chemotherapy which includes the following drugs: etoposide (E), prednisone (P), vincristine (O), cyclophosphamide (C), doxorubicin (H), and rituximab (R). The drug campath will be given by IV infusion on the first day of treatment over several hours. When this infusion is completed, the drug rituximab will be given by IV infusion over several hours. When the rituximab IV infusion is complete, the drugs doxorubicin, etoposide, and vincristine will each be given by continuous IV infusion over the next 4 days (that is, continuously for a total of 96 hours). Cyclophosphamide will be given by IV infusion on Day 5 after you have received the previous chemotherapy drugs. Prednisone will be given by mouth (orally) twice each day for 5 days. You will take the first dose of prednisone 8-12 hours before starting the campath.

You will receive the drug filgrastim by subcutaneous (under the skin) injection starting on Day 6 to increase white blood cell counts. Filgrastim will be continued until your white blood counts have reached acceptable levels. The dose of doxorubicin, etoposide, and/or cyclophosphamide may be "adjusted" up or down depending on your white blood cell count. You will be given a drug commonly known as Bactrim to be taken by mouth (orally) three times a week (for example, on a Monday-Wednesday-Friday schedule) to guard against possible infections. You will receive a drug called fluconazole to prevent fungal infections, and a drug called acyclovir to prevent certain viral infections. You will also receive a drug each day to be taken by mouth (orally) to guard against stomach ulcers, such as omeprazole. In addition, you will receive colace, or equivalent, by mouth twice daily to prevent constipation. If constipation becomes severe, you may also receive the laxative known as lactulose.

The EPOCH-RC therapy will be repeated every twenty-one (21) days, which is known as a "cycle" of therapy, for a total of 6 cycles. Following the fourth and sixth treatment cycles (approximately weeks 12 and 18) of EPOCH-RC, your doctor will evaluate you with blood tests and CT/MRI scans.

MEDICAL RECORD

CONTINUATION SHEET for either:

NIH 2514-1, Consent to Participate in A Clinical Research Study

NIH 2514-2, Minor Patient's Assent to Participate In A Clinical Research

Study

STUDY NUMBER: 10-C-0011 CONTINUATION:  pages

#### **EPOCH-RC Treatment Schema**

| | Da | y of | Trea | atm | ent | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | 0 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 11 | 12 | 13 | <br>21* |
| Campath | | X | | | | | | | | | | | | | |
| Rituximab | | X | | | | | | | | | | | | | |
| Etoposide | | Х- | | _ | | $\rightarrow$ | | | | | | | | | |
| Prednisone | X | X | X | X | X | X | | | | | | | | | |
| Vincristine | | Х- | | | | $\rightarrow$ | | | | | | | | | |
| Cyclophosphamide | | | | | | X | | | | | | | | | |
| Doxorubicin | | X – | | | | $\rightarrow$ | | | | | | | | | |
| Filgrastim | | | | | | | X* | * | <del></del> | | | | | | |

<sup>\*</sup> This twenty-one day (21) period will be known as a "cycle" of therapy. Therapy will be repeated for a total of 6 cycles. During the course of treatment, you may also receive the following drugs: Bactrim, fluconazole, acyclovir, omeprazole, and colace. On the first cycle of therapy the start of rituximab and EPOCH chemotherapy may be delayed until the following day if toxicity during the campath infusion caused a prolonged infusion time.

Research tests: We would like to perform research studies on your blood and tumor tissue to look at different genes and proteins that may be involved in the development of your lymphoma or the reaction of the immune system. We will not examine mutations of genes from your normal tissue without obtaining additional permission from you. We plan to do a tissue biopsy before you start treatment and after the first cycle of therapy. Biopsies of tumor will be done with local or general anesthesia. The tumor biopsies are being performed for two reasons; first to confirm your diagnosis and second to perform research tests on the tumor. These biopsies will give us important information about your tumor. Biopsies requiring major surgery (opening the chest or abdomen) will only be done if necessary for medical care and will not be done for experimental purposes. It is important, however, for you to understand that in some cases, biopsies of tumor may be done primarily for experimental purposes. These biopsies are optional for participation in the study but are important to help us learn how to better treat diffuse large B-cell and Hodgkin lymphomas.

<sup>\*\*</sup> Filgrastim will continue to be given to you until your blood counts have reached acceptable levels.

| Study | MEDICAL RECORD | CONTINUATION SHEET for either: NIH 2514-1, Consent to Participate in A Clinical Research Study NIH 2514-2, Minor Patient's Assent to Participate In A Clinical Research Study |
|---|---|---|
|---|---|---|

STUDY NUMBER: 10-C-0011 CONTINUATION:  pages

# **Optional Post Cycle 1 Biopsy**

The biopsy to be performed is exclusively for research purposes and will not benefit you. It might help other people in the future.

# When you are finished taking the drugs (treatment)

If all evidence of disease has disappeared, we will schedule periodic visits to the Clinical Center for follow-up examination and tests. If the disease does not disappear entirely or if it should recur after having disappeared for a period of time, then you may need further therapy. At that time, you will be given the opportunity of participating in additional research protocols that may be appropriate for you. If no such protocols are available, you will be returned to the care of your local physician. We will continue to contact you and/or your local physician to see how you are doing even after you have completed treatment on this protocol. It is important to stress that participation in this protocol does not mean you will receive long-term medical care here at the Clinical Center.

#### **Birth Control**

If you are a woman who is breast feeding or pregnant, you may not take part in the study because we don't know how this medicine would affect your baby or your unborn child. If you are a woman who can become pregnant, or are the partner of a woman who can become pregnant, you will need to practice an effective form of birth control before starting study treatment, during study treatment, and for 24 months after you finish study treatment. If you think that you or your partner is pregnant, you should tell your study doctor or nurse at once. For male subjects, you should practice contraception for the duration of the study and 12 months after completion of treatment.

Effective forms of birth control include:

- abstinence
- intrauterine device (IUD)
- hormonal [birth control pills, injections, or implants]
- tubal ligation
- vasectomy

# **Risks or Discomforts of Participation**

# What side effects or risks can I expect from being in this study?

# Risks associated with procedures

The risks associated with bone marrow biopsies are pain, bleeding and local infection. Risks of tissue biopsies include pain, bleeding, infection, and the risks to the particular area undergoing surgery. A biopsy of tumor may require general anesthesia but only for the purpose of making a diagnosis. General anesthesia will not be performed to obtain biopsies for research purposes.

| MEDICAL RECORD | CONTINUATION SHEET for either: NIH 2514-1, Consent to Participate in A Clinical Research Study NIH 2514-2, Minor Patient's Assent to Participate In A Clinical Research Study |
|---|---|
| | Study |

STUDY NUMBER: 10-C-0011 CONTINUATION:  pages

General anesthesia itself is generally very safe but has a very small risk of major complications such as heart attack or stroke. The surgical and anesthetic risks will be explained to you in more detail at the time of surgery, if this is needed.

You may be required to undergo a lumbar puncture if indicated. A small amount of spinal fluid (about 1-2 teaspoons) is removed and will be tested for the presence of lymphoma cells. A lumbar puncture is done by inserting a small sterile needle through the skin and muscle, going between the bones of the spine in the lower back until the needle punctures the spinal canal covering. The spinal fluid will then drain out through the needle on its own.

In order to receive this treatment, you will need to have a central venous catheter. This is catheter is placed under the skin of the chest wall and enters a major vein in the chest. There are several types of catheters including those which must be removed after each cycle of chemotherapy (temporary type) and those which may be kept for the duration of therapy (permanent type). These options will be discussed with you. The risks associated with placing some catheters include pain, bleeding, infection and collapsed lung. The long term risks of the catheter include infection, and clotting of your veins. If these occur, it may be necessary to remove the catheter. These risks will be explained to you in more detail at the time of insertion.

You may have side effects while on the study. Every one taking part in the study will be watched carefully for any side effects. However, doctors don't know all the side effects that may happen. Side effects may be mild or serious. Your health care team may give you medicines to help lessen side effects. In some cases, side effects can be serious or long-lasting or may never go away. There is also the risk of death from either the treatment or your disease.

You should talk to your doctor about any side effects that you have while taking part in the study.

Most of the side effects related to the treatment are listed in this form, but they will vary from person to person. There may be other side effects that we don't know about.

# **Side Effects of Campath**

**Likely:** These side effects occur in greater than 50% of patients

- Mild flu-like symptoms such as chills, fever (usually occur only with the first dose and decreased or absent with each following dose). Stopping or increasing the time it takes to give you campath may make these side effects go away.
- Decreased white blood cells (including normal T-cells), which may increase the risk of infection (bacterial, viral, fungal, parasitic); you will be given medicines to prevent infections.
- Decreased red blood cells (anemia), which may make you feel more easily tired, or even out of breath when performing simple daily tasks. It may also cause you to feel lightheaded, or have a rapid heartbeat. If you become symptomatic, red blood cell transfusion may be needed.

PATIENT IDENTIFICATION

#### **CONTINUATION SHEET for either:**

NIH-2514-1 (07-09) NIH-2514-2 (10-84) P.A.: 09-25-0099

| MEDICAL RECORD | CONTINUATION SHEET for either: NIH 2514-1, Consent to Participate in A Clinical Research Study NIH 2514-2, Minor Patient's Assent to Participate In A Clinical Research Study |
|---|---|
|---|---|

STUDY NUMBER: 10-C-0011 CONTINUATION:  pages

- Decreased platelet counts, which may increase the risk of bleeding or bruising. If bleeding becomes serious such bleeding from the gastro-intestinal tract, platelet transfusion will be warranted.
- Asymptomatic virus infection, in particular a virus called cytomegalovirus (CMV). CMV is a common virus that infects most people worldwide. It is a member of the herpesvirus family. Other members of the herpesvirus family cause chickenpox, infectious mononucleosis, fever blisters, and genital herpes. These viruses all share the ability to remain alive, but dormant, in the body for life. The virus lives in the body silently without causing obvious damage or illness but may reactivate when the immune system weakens. Even upon reactivation, there are usually no symptoms produced and is detected only on a blood test. You will be monitored closely with a blood test each time you return to clinic for signs of this infection.

**Less likely**: These side effects occur in 10-50% of patients:

These usually occur only with the first dose and are decreased or absent with each following dose.

- Skin rash
- itching
- Nausea
- Vomiting
- diarrhea
- general sick feeling
- decreased appetite
- headache
- fatigue
- low or high blood pressure
- shortness of breath
- cough
- rapid heart beat
- sweating
- muscle pain
- sepsis increased risk of bacterial and fungal infections

**Occasional:** These side effects occur in <10% of patients:

- dizziness
- dysesthesia or paresthesia (abnormal touch sensation)
- tremors
- insomnia
- sweating
- abnormal taste
- vasodilatation (increased blood flow)

PATIENT IDENTIFICATION

CONTINUATION SHEET for either:

NIH-2514-1 (07-09)

NIH-2514-2 (10-84)

P.A.: 09-25-0099

File in Section 4: Protocol Consent

| MEDICAL RECORD | CONTINUATION SHEET for either: NIH 2514-1, Consent to Participate in A Clinical Research Study NIH 2514-2, Minor Patient's Assent to Participate In A Clinical Research Study |
|---|---|
|---|---|

STUDY NUMBER: 10-C-0011 CONTINUATION:  pages

- confusion
- anxiety
- constipation
- leg edema

**Unlikely:** These side effects occur in <1% of patients.

- joint pain
- conjunctivitis
- deep vein thrombosis

Unlikely, but serious: These side effects are severe, life threatening, or cause death.

- Allergic reactions with any of the following symptoms:
- Marked lowering of the blood pressure, throat tightness, shortness of breath, severe skin rash
- Development of other cancers or recurrence of a past cancer.
- Heart rhythm, kidney, and lung problems caused by chemicals released into your blood from dead cancer cells; you will receive extra fluids before you start your treatment with campath to flush any extra chemicals out of your body, and you will also be given medicine to help control the chemical balance of your blood.
- Serious viral infection
- Changes in liver enzymes
- Cardiac arrhythmias
- Seizure
- Leukoencephalopathy Progressive loss of neurological function, the most prominent symptoms are clumsiness, progressive weakness, visual, speech and sometimes personality changes
- Abnormal clotting of the blood resulting in serious complications such clotting of blood vessels in the lungs.

Since campath can cause a prolonged lowering of lymphocytes (white blood cells), you may develop an increased risk for serious infections, the development of other tumors, or the recurrence of a previous cancer. Also, it is important to know that patients may develop other unexpected side effects and these could lead to serious organ damage or even death.

#### **Side Effects of EPOCH-R:**

#### Likely:

- Lowered white blood cell count that may lead to infection.
- Lowered platelets which may lead to an increase in bruising or bleeding.
- Lowered red blood cells which may cause anemia, tiredness, or shortness of breath.
- Should low counts occur, they can be treated with blood products (transfusions), antibiotics, and there may be a reduction in the amount of drug given to you.
- Constipation.
- Fatigue or tiredness

| • rangue of thedness. | |
|------------------------|-------------------------------------|
| PATIENT IDENTIFICATION | CONTINUATION SHEET for either: |
| | NIH-2514-1 (07-09) |
| | NIH-2514-2 (10-84) |
| | P.A.: 09-25-0099 |
| | File in Section 4: Protocol Consent |

| MEDICAL RECORD | CONTINUATION SHEET for either: NIH 2514-1, Consent to Participate in A Clinical Research Study NIH 2514-2, Minor Patient's Assent to Participate In A Clinical Research |
|---|---|
| | Study |

STUDY NUMBER: 10-C-0011 CONTINUATION:  pages

- Tingling of fingers and/or toes.
- Hair loss.
- Fever and/or chills.
- Time away from work.
- Urine colored red for a day or two after the doxorubicin infusion.
- Fingernail and toenail changes.
- Tearing or dry eyes.
- Runny nose.
- Bony pain.

#### Less Likely:

- Nausea and/or vomiting.
- Loss of appetite, change in taste and weight loss.
- Temporary shortness of breath or dizziness while receiving rituximab.
- Headaches.
- Muscle aches and muscle weakness.
- Hoarseness or pain in the jaw.
- Elevated blood sugar levels.
- Elevated or decreased blood pressure.
- Confusion.
- Mouth & throat sores. Temporary irritation to the mouth may lead to mouth ulcers (similar to canker sores). Medications to numb the mouth may ease the mouth discomfort.
- Stomach ulcers.
- Skin rashes and/or dry skin.
- Loss of control of muscles or reflexes.
- Abnormalities in blood results such as elevated liver enzymes, low blood protein and low blood calcium.
- Mood changes such as agitation or depression.
- Trouble sleeping.

#### Rare, But Serious:

- Severe constipation may result in abdominal pain and cramping.
- Bladder irritation with painful and bloody urine.
- Damage to the heart muscle.
- Skin rash that may be serious and life-threatening.
- Allergic reaction that may be severe or life-threatening. Symptoms may include difficulty breathing, low blood pressure, fast heart rate, and sweating.
- Severe hepatitis (liver infection) in those patients who are carriers of the hepatitis virus. Patients who may have had prior exposure to the hepatitis B and C virus may be at an increased risk of recurrence of the virus that may lead to severe liver damage that can be life-threatening. You doctor will screen you for the hepatitis virus before beginning

# PATIENT IDENTIFICATION CONTINUATION SHEET for either: NIH-2514-1 (07-09) NIH-2514-2 (10-84) P.A.: 09-25-0099 File in Section 4: Protocol Consent

| MEDICAL RECORD | CONTINUATION SHEET for either: NIH 2514-1, Consent to Participate in A Clinical Research Study NIH 2514-2, Minor Patient's Assent to Participate In A Clinical Research |
|---|---|
| | Study |

STUDY NUMBER: 10-C-0011 CONTINUATION:  pages

treatment on this study. If you test positive for the virus, you will be closely monitored for signs of the infection, and you will be treated, if appropriate, by your doctor.

#### **Reproductive risks:**

Many of the drugs used in this treatment program are toxic to the cells in the ovary and testicle and may produce sterility. Recovery of normal fertility is not well studied although we know that some patients treated with this combination have remained fertile after the therapy has been completed. For this reason, men who are about to receive this treatment should, if they wish to have children in the future, consider sperm banking before start of the treatment.

# **Potential Benefits of Participation**

# Are there benefits to taking part in this study?

It is likely that most patients will have at least a temporary improvement from treatment with Campath and EPOCH-R chemotherapy. However, we cannot be certain if you will be cured of your lymphoma and it is possible that you may not respond to treatment.

In addition, your participation in this protocol may contribute to advances in the understanding of and treatment for your disease

#### **Alternative Approaches or Treatments**

# What other choices do I have if I do not take part in this study?

We do not know at this point whether the combination of drugs we are offering to you is more effective, less effective or the same as the standard combination chemotherapy for your disease.

Instead of being in this study, you have these options:

- Other combination drug regimens and other schedules of the same drugs used in this study. For example, a chemotherapy called R-ICE given in the conventional manner would be suitable standard therapy for your condition. This is given either by itself or as a bridge to stem-cell transplant.
- Treatment with single drugs. This is known to produce brief responses of a few months'
  duration in many patients but to have little beneficial effect in long-term control of the
  disease
- Radiation (X-ray) treatments. This can stop tumor growth in particular locations, such as bone, abdomen, and other sites but is not successful in controlling the disease overall unless the disease is very localized at the start of therapy.
- Surgery. As with radiation, surgery can be successful in removing tumor from particular locations but cannot be used successfully to remove all lymphoma cells from the body, since the disease is almost always present in multiple locations. Also, surgery cannot be used against tumor in some of the organs most commonly involved by lymphoma, such as the liver or the lungs

# PATIENT IDENTIFICATION CONTINUATION SHEET for either:

NIH-2514-1 (07-09) NIH-2514-2 (10-84)

P.A.: 09-25-0099

| MEDICAL RECORD | CONTINUATION SHEET for either: NIH 2514-1, Consent to Participate in A Clinical Research Study NIH 2514-2, Minor Patient's Assent to Participate In A Clinical Research |
|---|---|
| | Study |

STUDY NUMBER: 10-C-0011 CONTINUATION:  pages

- Waiting, without active therapy. Although a period of watchful waiting is appropriate treatment for some kinds of tumors, in lymphomas similar to yours, the disease will often grow and spread rapidly if no treatment is administered.
- Getting treatment or care for your cancer without being in a study
- Taking part in another study
- Getting comfort care, also called palliative care. This type of care helps reduce pain, tiredness, appetite problems and other problems caused by the cancer. It does not treat the cancer directly. Instead, it tries to improve how you feel. Comfort care tries to keep you as active and comfortable as possible.

Please talk to your doctor about these and other options.

# **Stopping Therapy**

Your doctor may decide to stop your therapy for the following reasons:

- if he/she believes that it is in your best interest
- if your disease comes back during treatment
- if you have side effects from the treatment that your doctor thinks are too severe
- if new information shows that another treatment would be better for you

In this case, you will be informed of the reason therapy is being stopped.

You can stop taking part in the study at any time. However, if you decide to stop taking part in the study, we would like you to talk to the study doctor and your regular doctor first.

If you decide at any time to withdraw your consent to participate in the trial, we will not collect any additional medical information about you. However, according to FDA guidelines, information collected on you up to that point may still be provided to designated representatives. If you withdraw your consent and leave the trial, any samples of yours that have been obtained for the study and stored at the NCI can be destroyed upon request. However, any samples and data generated from the samples that have already been distributed to other researchers or placed in the research databases can**not** be recalled and destroyed.

#### Research Subject's Rights

Participation in this investigational treatment protocol is voluntary; you may discontinue your participation in the protocol at any time. You will be given a copy of the consent for your records. There are no penalties imposed for withdrawing from the protocol. Patients may ask questions of the staff, and indeed are encouraged to do so. Any significant new findings that relate to your treatment will be discussed with you. It is possible that participation in this study may make you ineligible to participate in other research studies, which limit the type or number of prior treatments patients may have received.

#### PATIENT IDENTIFICATION CONTINUATION SHEET for either:

NIH-2514-1 (07-09) NIH-2514-2 (10-84)

P.A.: 09-25-0099

| MEDICAL RECORD | CONTINUATION SHEET for either: NIH 2514-1, Consent to Participate in A Clinical Research Study NIH 2514-2, Minor Patient's Assent to Participate In A Clinical Research Study |
|---|---|
| | 2 |

STUDY NUMBER: 10-C-0011 CONTINUATION:  pages

# What are the costs of taking part in this study?

If you choose to take part in the study, the following will apply, in keeping with the NIH policy:

- You will receive study treatment at no charge to you. This may include surgery, medicines, laboratory testing, x-rays or scans done at the Clinical Center, National Institutes of Health (NIH), or arranged for you by the research team to be done outside the Clinical Center, NIH if the study related treatment is not available at the NIH.
- There are limited funds available to cover the cost of some tests and procedures performed outside the Clinical Center, NIH. You may have to pay for these costs if they are not covered by your insurance company.
- Medicines that are not part of the study treatment will not be provided or paid for by the Clinical Center, NIH.
- Once you have completed taking part in the study, medical care will no longer be provided by the Clinical Center, NIH.

# Will your medical information be kept private?

We will do our best to make sure that the personal information in your medical record will be kept private. However, we cannot guarantee total privacy. Organizations that may look at and/or copy your medical records for research, quality assurance, and data analysis include:

- The National Cancer Institute (NCI) and other government agencies, like the Food and Drug Administration (FDA), which are involved in keeping research safe for people.
- National Cancer Institute Institutional Review Board

A description of this clinical trial will be available on <a href="http://www.Clinicaltrials.gov">http://www.Clinicaltrials.gov</a>, as required by U.S. Law. This Web site will not include information that can identify you. At most the Web site will include a summary of the results. You can search this Web site at any time.

# **Certificate of Confidentiality**

To help us protect your privacy, we have obtained a Certificate of Confidentiality. The researchers can use this Certificate to legally refuse to disclose information that may identify you in any federal, state, or local civil, criminal, administrative, legislative, or other proceedings, for example, if there is a court subpoena. The researchers will use the Certificate to resist any demands for information that would identify you, except as explained below.

You should also know that there are several circumstances in which the Certificate does not provide coverage. These include when information:

- will be used for auditing or program evaluation internally by the NIH; or
- must be disclosed to meet the legal requirements of the federal Food and Drug Administration (FDA).

| PATIENT IDENTIFICATION | CONTINUATION SHEET for either: |
|------------------------|-------------------------------------|
| | NIH-2514-1 (07-09) |
| | NIH-2514-2 (10-84) |
| | P.A.: 09-25-0099 |
| | File in Section 4: Protocol Consent |

| MEDICAL RECORD | CONTINUATION SHEET for either: NIH 2514-1, Consent to Participate in A Clinical Research Study NIH 2514-2, Minor Patient's Assent to Participate In A Clinical Research Study |
|---|---|
|---|---|

STUDY NUMBER: 10-C-0011 CONTINUATION:  pages

- is necessary for your medical treatment and you have consented to this disclosure;
- is for other research.

In addition, identifiable, sensitive information protected by this Certificate cannot be admissible as evidence or used for any purpose in any action, suit, or proceeding without your consent.

You should understand that a Certificate of Confidentiality does not prevent you or a member of your family from voluntarily releasing information about yourself or your involvement in this research. If an insurer, employer, or other person obtains your written consent to receive research information, then the researchers will not use the Certificate to withhold that information.

The Certificate of Confidentiality will not protect against the required reporting by hospital staff of information on suspected child abuse, reportable communicable diseases, and/or possible threat of harm to self or others.

#### **Conflict of Interest**

The National Institutes of Health (NIH) reviews NIH staff researchers at least yearly for conflicts of interest. This process is detailed in a Protocol Review Guide. You may ask your research team for a copy of the Protocol Review Guide or for more information. Members of the research team who do not work for NIH are expected to follow these guidelines but they do not need to report their personal finances to the NIH.

Members of the research team working on this study may have up to \$15,000 of stock in the companies that make products used in this study. This is allowed under federal rules and is not a conflict of interest.

#### **Optional Biopsy**

The biopsy to be performed is exclusively for research purposes and will not benefit you. It might help other people in the future.

If you agree to have the optional biopsy, you will be asked to sign a separate procedure consent before you have the procedure.

#### **Use of Specimens and Data for Future Research**

To advance science, it is helpful for researchers to share information they get from studying human samples. They do this by putting it into one or more scientific databases, where it is stored along with information from other studies. A researcher who wants to study the information must apply to the database and be approved. Researchers use specimens and data stored in scientific databases to advance science and learn about health and disease.

We plan to keep some of your specimens and data that we collect, use them for future research and share them with other researchers. We will not contact you to ask about each of these future uses. These specimens and data will be stripped of identifiers such as name, address or account number, so that they may be used for future research on any topic and shared broadly for

NIH-2514-1 (07-09) NIH-2514-2 (10-84) P.A.: 09-25-0099

| MEDICAL RECORD | CONTINUATION SHEET for either: NIH 2514-1, Consent to Participate in A Clinical Research Study NIH 2514-2, Minor Patient's Assent to Participate In A Clinical Research |
|---|---|
| | Study |

STUDY NUMBER: 10-C-0011 CONTINUATION:  pages

research purposes. Your specimens and data will be used for research purposes only and will not benefit you. It is also possible that the stored specimens and data may never be used.

Results of research done on your specimens and data will not be available to you or your doctor. It might help people who have cancer and other diseases in the future. If you do not want your stored specimens and data used for future research, please contact us in writing and let us know that you do not want us to use your specimens and data. Then any specimens that have not already been used or shared will be destroyed and your data will not be used for future research. However, it may not be possible to withdraw or delete materials or data once they have been shared with other researchers.

NIH-2514-1 (07-09) NIH-2514-2 (10-84) P.A.: 09-25-0099

MEDICAL RECORD

#### CONSENT TO PARTICIPATE IN A CLINICAL RESEARCH STUDY

Adult Patient or

• Parent, for Minor Patient

STUDY NUMBER: 10-C-0011

CONTINUATION:  pages

#### OTHER PERTINENT INFORMATION

1. Confidentiality. When results of an NIH research study are reported in medical journals or at scientific meetings, the people who take part are not named and identified. In most cases, the NIH will not release any information about your research involvement without your written permission. However, if you sign a release of information form, for example, for an insurance company, the NIH will give the insurance company information from your medical record. This information might affect (either favorably or unfavorably) the willingness of the insurance company to sell you insurance.

The Federal Privacy Act protects the confidentiality of your NIH medical records. However, you should know that the Act allows release of some information from your medical record without your permission, for example, if it is required by the Food and Drug Administration (FDA), members of Congress, law enforcement officials, or authorized hospital accreditation organizations.

- 2. Policy Regarding Research-Related Injuries. The Clinical Center will provide short-term medical care for any injury resulting from your participation in research here. In general, no long-term medical care or financial compensation for research-related injuries will be provided by the National Institutes of Health, the Clinical Center, or the Federal Government. However, you have the right to pursue legal remedy if you believe that your injury justifies such action.
- **3. Payments.** The amount of payment to research volunteers is guided by the National Institutes of Health policies. In general, patients are not paid for taking part in research studies at the National Institutes of Health. Reimbursement of travel and subsistence will be offered consistent with NIH guidelines.
- 4. **Problems or Questions.** If you have any problems or questions about this study, or about your rights as a research participant, or about any research-related injury, contact the Principal Investigator, Wyndham Wilson, M.D., Ph.D.; Building 10, Room 4N115, Telephone: 240-760-6092. You may also call the Clinical Center Patient Representative at 301-496-2626. If you have any questions about the use of your specimens or data for future research studies, you may also contact the Office of the Clinical Director, Telephone: 240-760-6070.
- 5. Consent Document. Please keep a copy of this document in case you want to read it again.

PATIENT IDENTIFICATION

CONSENT TO PARTICIPATE IN A CLINICAL RESEARCH STUDY (Continuation Sheet)

• Adult Patient or

Parent, for Minor Patient

NIH-2514-1 (07-09) P.A.: 09-25-0099

MEDICAL RECORD

# CONSENT TO PARTICIPATE IN A CLINICAL RESEARCH STUDY

• Adult Patient or

• Parent, for Minor Patient

STUDY NUMBER: 10-C-0011

CONTINUATION:  pages

| COMPLETE APPROPRIATE ITEM(S) BELOW: | | | |
|---|---|---|---|
| A. Adult Patient's Consent | | <b>B.</b> Parent's Permission for Minor Patient. | |
| I have read the explanation about | this study | I have read the explanation about this study | |
| and have been given the opportun | ity to | and have been given the opportunity to | |
| discuss it and to ask questions. Il | nereby | discuss it and to ask questions. I hereby give | |
| consent to take part in this study. | | permission for my child to take part in this | |
| | | study. | |
| | | (Attach NIH 2514-2, Minor's A | ssent, if |
| | | applicable.) | |
| Signature of Adult Patient/ | Date | Signature of Parent(s)/ | Date |
| Legal Representative | | Guardian | |
| | _ | | |
| Print Name | | Print Name | |
| C. Child's Verbal Assent (If Ap | plicable) | | |
| The information in the above co | onsent was d | lescribed to my child and my cl | nild agrees to |
| participate in the study. | | | |
| Signature of Parent(s)/Guardian | Date | Print Name | |
| THIS CONSENT DO | CUMENT H | IAS BEEN APPROVED FOR U | SE |
| FROM SEPTEMBER 24, 2018 THROUGH OCTOBER 15, 2019. | | | |
| Signature of Investigator | Date | Signature of Witness | Date |
| Print Name | | Print Name | |
| FIIII INAIIIC | | FIIII INAIIIE | |

PATIENT IDENTIFICATION

# CONSENT TO PARTICIPATE IN A CLINICAL RESEARCH STUDY (Continuation Sheet)

• Adult Patient or NIH-2514-1 (07-09)

• Parent, for Minor Patient

P.A.: 09-25-0099